CLINICAL TRIAL: NCT05583942
Title: A Pilot Randomized Clinical Trial of Transcutaneous Auricular Vagus Nerve Stimulation for the Treatment of Steroid Resistant Nephrotic Syndrome in Children
Brief Title: A Pilot Trial of taVNS for SRNS in Children (kidNEY-VNS)
Acronym: kidNEY-VNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-0488-A; 1R01DK131091-01A1 (NIH)
Record Dates: First submitted 2022-09-26; First posted 2022-10-18 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Nephrotic Syndrome in Children; Minimal Change Disease; Focal Segmental Glomerulosclerosis
Keywords: vagus nerve stimulation; pediatric; nephrology
MeSH Terms: conditions — Nephrosis, Lipoid; Glomerulosclerosis, Focal Segmental

STUDY DESIGN:
Intervention Model Description: Randomized double blind sham controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be double-blinded to the investigators and participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group (Experimental): The intensity setting for pulse amplitude will be adjusted to the participant's tolerance (if a sensation is felt) to a maximum level of 3.
  Interventions: Device: trascutaneous auricular vagus nerve stimulation
- Sham Group (Sham Comparator): The sham device will be altered internally so that electrical stimulation is not delivered, but the device will appear to function. Externally, the sham device will look identical to the taVNS device. The participant will be told to increase the intensity until tolerated if a sensation is felt, but will be asked to stop at a maximum level of 3.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: trascutaneous auricular vagus nerve stimulation — The device to be used is the Roscoe Medical TENS 7000, a commercially available handheld electrical pulse generator, and an ear clip to be placed at the left ear for stimulation. Custom-made ear clips with electrode gel will be placed near the entrance to the canal of the ear to provide stimulation to the auricular branch. The handheld electrical pulse generator will be programmed to deliver electrical stimulation pulses to the cymba concha stimulating the auricular branch of the vagus nerve.
  Other Names: Roscoe TENS 7000
  Arms: Intervention Group
Device: Sham device — The device will appear to function but no electrical stimulation will be delivered.
  Other Names: Roscoe TENS 7000
  Arms: Sham Group

SUMMARY:
Children with steroid resistant nephrotic syndrome (SRNS) are exposed to prolonged courses of immunosuppressant medications. Given the adverse side effect profiles and variable efficacy of these medications, there is an urgent need to identify novel and safe therapies to treat nephrotic syndrome in children. Stimulation of the vagus nerve, which can be activated noninvasively by transcutaneous auricular vagus nerve stimulation (taVNS), has immunomodulatory effects mediated by the inflammatory reflex and spleen. taVNS has become a therapy of interest for treating chronic immune mediated illnesses. The aims of the study are (1) To determine the feasibility of protocol implementation and tolerability of taVNS in the treatment of nephrotic syndrome in children (2) To establish proof-of-concept and generate statistical estimates of variance parameters and effect sizes for treatment response outcomes in children with nephrotic syndrome randomized to taVNS therapy compared with sham therapy (3) To investigate the effects of taVNS on inflammatory markers in children with nephrotic syndrome.

DETAILED DESCRIPTION:
A parallel, double blinded, randomized placebo controlled trial comparing daily taVNS use with sham therapy will be conducted in children 3 to 17 years of age with SRNS. Ten participants with SRNS, defined as lack of response to steroids after 4 weeks, will be randomized 1 to 1 to taVNS or sham therapy. Participants will be enrolled at two pediatric tertiary hospitals over a two year time period, with completion of the study by year three. All participants will perform daily taVNS therapy (active for taVNS arm or inactive for sham arm) for 5 minutes each day for a total of 26 weeks.

Participants will monitor heart rate with each treatment and log home urine results. Participants will be monitored monthly with in person study visits at Weeks 8, 16 and 26 alternating with virtual telehealth visits at Weeks 4, 12 and 20. Biosample specimens will be collected at baseline, 8 weeks, 16 weeks and 26 weeks. There will be a follow up period of an additional 26 weeks. All participants will be given the option to receive the active taVNS treatment at the end of the randomized period.

Study Phases The study will consist of three parts. Part 1 - Screening Period- up to 8 weeks. Informed consent/assent will be obtained at screening prior to the conduct of any study-related procedures. Participants will be screened to confirm inclusion/exclusion criteria are met. Participants must be off steroid treatment for 14 days prior to Day 1 and the participant must be in remission (negative UPC on first morning urine) on Day 1.

Part 2 - Randomized Control Period - 26 weeks: Thirty participants with FRNS who meet all of the eligibility criteria will be randomized 1:1 to either taVNS or sham treatment. A trainer will instruct the parent/guardian on use of the device at the randomization visit. Participants will use the intervention device as directed for 5 minutes per day for 26 weeks. Participants will be monitored monthly with in-person study visits at Weeks 8, 16 and 26 alternating with virtual remote video visits at Weeks 4, 12 and 20. The visit window will be +/- 7 days. At each in person visit, we will conduct:

* Vital signs and physical examination
* Assessment for nephrotic syndrome relapses. Home urine protein logs will be reviewed.
* Blood and urine samples will be collected at each in person visit.
* Assessment of study intervention adherence. Parents/guardians will meet with the trainer and will be reoriented on taVNS device use at each visit as a safety measure. The device counter number will be recorded as a measure of adherence.
* Monitor for adverse events and tolerability: Parents/guardians will share a study log with investigators, which describes daily taVNS use, side effects, and any changes in heart rate.

At each virtual remote video visit, we will observe the participant while doing the intervention procedure, assess for nephrotic syndrome relapses, and monitor for any adverse events.

Part 3 - Follow Up Period - 26 weeks: At the completion of the randomized period, participants will be followed for an additional 26 weeks to assess clinical status. For those who stop the intervention, study visits will occur in-person during regularly scheduled clinical visits or via telehealth visit every 8 weeks, whichever is sooner. Participants will be assessed for the number of nephrotic syndrome relapses and home urine protein logs will be reviewed. First morning UPC will be recorded. All participants will be given the option to receive the active taVNS treatment at the end of the randomized period. Unblinding of treatment assignment from the randomized phase will not occur prior to consent for open-label use. As open-label extension trials may introduce significant bias, data obtained from these participants will not be considered part of this research and no statistical analysis will be carried out. However, clinical status and safety will continue to be monitored. In person study visits will occur every 8 weeks for those continuing use of taVNS.

ELIGIBILITY:
Inclusion Criteria:

* Steroid Resistant Nephrotic Syndrome- defined as lack of remission after 4 weeks of therapy of prednisolone/prednisone at standard dose1
* Age 3-17 years
* eGFR ≥30 ml/min/1.73 m2 (by modified Schwartz formula)
* MCD or FSGS diagnosis (per biopsy)
* Urine protein:creatinine (UPC) greater than 1.0
* Stable immunosuppression and ACE inhibitor/angiotensin receptor blocker treatment regimen for at least three months
* Evidence of B cell repletion for those exposed to rituximab
* Informed consent from the parent or guardian and assent from a minor of ≥ 7 years
* Ability to comply with the study protocol, in the investigator's judgment

Exclusion Criteria:

* Secondary causes of nephrotic syndrome (e.g. genetic, congenital, infectious)
* Steroid sensitive nephrotic syndrome
* History of genetic defects known to directly cause nephrotic syndrome (i.e., NPHS2 [podocin], NPHS1 [nephrin], PLCE1, WT1, or other known genetic cause)
* Any known inflammatory condition
* History of cardiac disease (arrhythmias, structural/functional abnormalities)
* Implantable electronic devices (pacemakers, defibrillators, hearing aids, cochlear implants or deep brain stimulators)
* Chronic rash or skin breakdown of the left ear at the cymba concha
* Pregnancy

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Success of Pilot Trial | Baseline to 26 weeks
  1. Unsuccessful: main study not practicable
     1. None of the primary feasibility and tolerability benchmarks are met, or
     2. One or more of the primary benchmarks are not met and there is low likelihood of reaching benchmarks even with protocol modifications or
     3. Serious adverse events related to the treatment.
  2. Probable Success: main study practicable with modifications to protocol. One or more of the primary benchmarks are not met, but there is a high likelihood that the benchmark can be met with protocol modifications.
  3. Successful: main study practicable without modifications. All of the primary benchmarks are met.

SECONDARY OUTCOMES:
Effect size for change in Change in quality of life (PedsQL) | Baseline to 26 weeks
  To calculate effect sizes for continuous main trial efficacy outcomes using a t test, Cohen's d test will be used.
Effect size for change in urine protein:creatinine | Baseline to 26 weeks
  To calculate effect sizes for continuous main trial efficacy outcomes using a t test, Cohen's d test will be used.
Effect size for change in lipid profile | Baseline to 26 weeks
  To calculate effect sizes for continuous main trial efficacy outcomes using a t test, Cohen's d test will be used.
Effect size for change in proportion with at least a 30 percent reduction in UPC | Baseline to 26 weeks
  To estimate effect sizes for dichotomous main trial efficacy outcomes using Fisher's exact test, odds ratios will be calculated outcomes using a t test, Cohen's d test will be used.
Recruitment rate | Baseline to 26 weeks
  Feasibility- %
Rate of completion of study | Baseline to 26 weeks
  Feasibility- %
Successful double-blinding | Baseline to 26 weeks
  Feasibility- %
Treatment adherence from home logs | Baseline to 26 weeks
  Feasibility- %
Adverse events | Baseline to 26 weeks
  Tolerability- %
Incidence of withdrawal due to adverse events | Baseline to 26 weeks
  Tolerability- %
Proof of Concept Decision Criteria | Baseline to 26 weeks
  A decision of whether to move forward with a larger trial will be made based on pre-determined proof of concept decision criteria. Once data from the two pilot trials are observed and collected, 1,000 bootstrap resamples with replacement will be carried out to construct the empirical 95% confidence interval (CI) for the relative risk.
Cytokines | Baseline to 26 weeks
  TNF, IL-6
Anti-nephrin antibodies | Baseline to 26 weeks
Whole blood monocyte stimulation test | 0 hours, 2 hours
  Change in monocyte cytokines at baseline and 2 hours post taVNS

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 12 months of study closure.
Access Criteria: Consent forms will be uploaded to clinical trials.gov. Data is available from the PI upon request.